CLINICAL TRIAL: NCT01273025
Title: Medicinal Effect of Lime Powder Regimen in HK-2 Cell Exposed to Lithogenic Crystals and Its Citraturic and Antioxidative Responses in Healthy Volunteers
Brief Title: Lime Powder Regimen in Healthy Volunteers
Acronym: LimePKphase1
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Chulalongkorn University (Other)
Responsible Party: Napatr Aungkasuvapala, Chulalongkorn University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PPK-10-003
Record Dates: First submitted 2011-01-05; First posted 2011-01-10 (Estimated); Last update posted 2011-01-10 (Estimated); Status verified 2011-01

CONDITIONS: Kidney Stone; Oxidative Stress
Keywords: pharmacokinetic; lime powder regimen; kidney stone; Oxidative stress
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Dietary Supplement: Lime powder regime — 1 sachet of lime powder regimen with 200 ml of water

SUMMARY:
The study aims to investigate the pharmacokinetic parameters and its antioxidative effects in Thai healthy men.

ELIGIBILITY:
Inclusion Criteria:

* Thai healthy male or female aged 18-45 years old
* BMI 18-25 kg/m2
* Normal medical history, physical examination and vital signs
* Normal screening laboratories
* no history of drug allergies
* Willingness to take part in the study and provide informed consent

Exclusion Criteria:

* History of GI, liver, kidney, allergic disease or any other disease that may interfere with the bioavailability of lime powder regimen
* History of alcohol or drug abuse
* Heavy smoking
* Receive any medication within 14 days prior to the study day

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2010-12; Primary Completion 2011-03 (Estimated); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
The pharmacokinetic parameters of plasma and urine citrate | 6 months
  The pharmacokinetic parameters of plasma and urine citrate incluiding Cmax, Tmax, Half life, AUC, and elimination rate constant

CONTACTS AND LOCATIONS:
Overall Officials: Poonsin Poungpairoj, BSc, Principal Investigator — Chulalongkorn University
Locations (1):
- Chula clinical research center, Bangkok, Thailand